CLINICAL TRIAL: NCT04937712
Title: Molecular Characterization and Cellular Infection Capacity of Urinary Viral Particles Isolated From SARS-CoV-2 and Association With Proximal Tubular Dysfunction, in Hospitalized Patients With COVID-19
Brief Title: Analysis of SARS-CoV2 Urine Viral Particles and Association With Proximal Tubular Dysfunction
Acronym: CovUrinePTD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Raphaël KORMANN, Principal investigator, Medical Doctor, Nephrologist, Central Hospital, Nancy, France
Other Study IDs: 2021-A00724-37
Record Dates: First submitted 2021-06-22; First posted 2021-06-24 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV2 Infection; Proximal Tubule Dysfunction
MeSH Terms: conditions — COVID-19 | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Reverse Transcriptase -Polymerase Chain Reaction (RT-PCR) for SARS-CoV2 in urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: RT-PCR SARS-COV2 in urine — proteinuria/renal phosphate leak/uricosuria/glycosuria/ aminoaciduria)
  Other Names: Proximal tubular dysfunction testing

SUMMARY:
The primary goal is to detect Severe Acute Respiratory Syndrome CoronaVirus 2 (SARS-CoV2) urine viral particles in patients in intensive care units, hospitalized for coronavirus Coronavirus Disease-19 (COVID-19) infection, and correlate the presence of the virus in the urine with proximal tubular dysfunction (defined by the association of at least 2 abnormalities: tubular proteinuria, renal phosphate leak, uricosuria, normoglycemic glycosuria, amino aciduria)

ELIGIBILITY:
Inclusion Criteria:

* Person and / or trustworthy person who has received complete information on the organization of the research and who has not opposed their participation and the use of their data
* Hospitalized for ≥ 48 hours and ≤ 10 days
* SARS-CoV-2 positive nasopharyngeal sample
* Severity criteria: Lung involvement described as compatible with SARS-CoV-2 on radiography or scanner and partial pressure of oxygne (PaO2) / Fraction of inspired oxygen (FiO2) ≤ 300 mmHg and / or respiratory rate (RR) ≥ 30 / min

Exclusion Criteria:

* Known chronic kidney disease, or initial Glomerular Filtration Rate (GFR) <60 ml / min / 1.73m2 or Renal Transplant
* Known proteinuria
* Known proximal tubulopathy
* Treatment with Forxiga

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in CHRU Nancy with severe SARS-CoV2 infection, with lung involvement.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV 2 viruria and its correlation with proximal tubule dysfunction | During the first 10 days of hospitalization
  Is the detection of viral particles in urine associated with proximal tubule dysfunction, defined by two or more of the following : proteinuria, phosphate leak, aminoaciduria, hyperuricuria, and/or glycosuria

SECONDARY OUTCOMES:
Capacity of infection of urine viral particles | During the first 10 days of hospitalization
  Study of the capacity for cell infection in vitro by viral particles detected in urine.
Sequencing viral particles to identify possible compartmentalization of the virus | During the first 10 days of hospitalization
  Study by sequencing of the compartmentalization of urinary and nasopharyngeal variants of SARS-CoV-2 in patients with positive urine for SARS-CoV-2.

CONTACTS AND LOCATIONS:
Locations (1):
- Chru Brabois, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kormann R, Jacquot A, Alla A, Corbel A, Koszutski M, Voirin P, Garcia Parrilla M, Bevilacqua S, Schvoerer E, Gueant JL, Namour F, Levy B, Frimat L, Oussalah A. Coronavirus disease 2019: acute Fanconi syndrome precedes acute kidney injury. Clin Kidney J. 2020 Jun 8;13(3):362-370. doi: 10.1093/ckj/sfaa109. eCollection 2020 Jun. PMID 32695327